CLINICAL TRIAL: NCT01646788
Title: Study of NMB Drug Ejecting Balloon for Arteriovenous Fistulae
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: N.M.B. Medical Applications Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NMB AVS HSR
Record Dates: First submitted 2012-07-16; First posted 2012-07-20 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Obstructive Lesions of Arteriovenous Dialysis Fistulae

ARMS (1):
- Experimental (Experimental): NMB's PTA Balloon catheter with Paclitaxel drug
  Interventions: Device: NMB Paclitaxel Drug Ejecting Balloon

INTERVENTIONS:
Device: NMB Paclitaxel Drug Ejecting Balloon — NMB's PTA Balloon catheter with drug

SUMMARY:
The purpose of this study is to demonstrate the safety and effectiveness of the use of NMB's percutaneous transluminal angioplasty (PTA) for the treatment of obstructive lesions of Arteriovenous (AV) Dialysis Fistulae/Grafts.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is 18 years old or older.
2. Native arteriovenous fistula or synthetic arteriovenous access graft performed/implanted more than 45 days before enrollment and at least one successful hemodialysis session performed.
3. Patient having obstructive lesion of native or synthetic arteriovenous dialysis fistulae/grafts, suitable for PTA procedure.
4. Patient who is willing and able to sign a written informed consent and that complies with procedures (including adherence to follow-up visits).

Exclusion Criteria:

1. Women who are pregnant or breast-feeding and women of childbearing potential who do not use adequate contraception.
2. Previous participation in another study with any investigational drug or device within the past 30 days.
3. Life expectancy of less than 12 months or factors making clinical and/or angiographic follow-up difficult.
4. Known hypersensitivity to paclitaxel or structurally-related compounds.
5. Severe reaction to contrast agents that cannot be adequately premedicated prior to procedure.
6. Stenosis with corresponding thrombosis treated within 7 days before enrollment.
7. Patient with known contraindications for aspirin or other anticoagulant/antiplatelet therapy.
8. Infected grafts/fistulae.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Restenosis rate | 6 months
  Binary Stenosis is defined as ≥50% narrowing in luminal diameter basen upon comparison with the adjacent normal vessel.
  Restenosis Rate - comparison shall be performed both to the patient previous data as well as to restenosis rate data published in the literature for standard PTA balloon catheter procedure

SECONDARY OUTCOMES:
restenosis rate | 1, 3 and 12 months
  As defined above in the primary end point
Easy insertion and removal | intraprocedural
Major adverse events rate | intraprocedural 1, 3, 6 and 12 months
  All adverse events will be reviewed by the Investigator and evaluated as follows:
  * Nature of the event.
  * Severity of the event - serious, moderate, mild.
  * Relation of the adverse event to the device - unrelated, possible, definite

CONTACTS AND LOCATIONS:
Locations (1):
- The Rabin Medical Center, Hasharon Hospital, Petah Tikva, Israel